CLINICAL TRIAL: NCT05524701
Title: The Effect of Short-term Sleep Restriction on Sweet and Fat Taste Preference and Perception.
Brief Title: Short-term Sleep Restriction on Taste Preference and Perception
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Professor Jason Gill, Professor, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200210063
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Sleep Restriction; Normal Sleep

STUDY DESIGN:
Intervention Model Description: A randomised crossover trial with one group undergoing two conditions- a sleep restriction condition and a normal sleep condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Restriction Condition (Experimental): Participants will be asked to restrict their sleep duration to a maximum of four hours per night (3 am to 7 am) for the two nights prior to the measurement day.
  Interventions: Behavioral: Sleep Restriction and Normal Sleep
- Normal Sleep Condition (Experimental): Participants will be asked to sleep for at least eight hours per night (11 pm to 7 am) for two nights prior to the measurement day.
  Interventions: Behavioral: Sleep Restriction and Normal Sleep

INTERVENTIONS:
Behavioral: Sleep Restriction and Normal Sleep — The intervention will consist of either sleep restriction (4 hours per night, 3 am to 7 am) or normal sleep (8 hours per night 11 pm to 7 am) for a duration of two nights.

SUMMARY:
The study aims is to investigate the effects of sleep restriction on sweet and fat taste perception and preference in both fasted and fed states. This is a randomised crossover trial with sleep restriction (4 hours per night for 2 nights) and normal sleep (at least 8 hours sleep for 2 nights) conditions, with a four-week washout period between conditions.

DETAILED DESCRIPTION:
Sleep restriction has been found to dysregulate appetite regulation, leading to an increased food intake, particularly of foods high in sugar and fat. It is unclear why sleep restriction leads to increased fat and sugar intake, but emerging evidence suggests that taste preference and perception may be influenced by the lack of sleep.

Sleep restriction leads to increased preference for sucrose. However it is unclear whether sleep restriction also alters perception of sweetness, or whether it affects preference or perception of dietary fat. It is also unclear, whether any changes in sweet and fat preference and perception due to sleep restriction differ between the fasted and fed states.

This study is a randomised crossover trial where each participant will undertake two conditions (sleep restriction and normal sleep) in a randomised order. In the sleep restriction condition, participants will be asked to restrict their sleep duration to a maximum of four hours per night for two nights, and in the normal sleep group they will be asked to sleep for at least eight hours per night for two nights. There will a 4-week wash-out period between conditions. After each condition (2 nights of normal sleep or 2 nights of sleep restriction), particpants asked to arrive in a fasted state for the assessments. They will initially undertake the Control of Eating Questionnaire (COEQ) and the Leeds Food Preference Questionnaire (LFPQ). Participants will then undertake the sweet and fat taste perception and preference tests (described below). Following this, all participants will be provided with a standardized breakfast meal, and 60 minutes later, the LFPQ and taste preference and perception tests will be repeated in fed state.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Self Reported sleep of >7 hours a night

Exclusion Criteria:

* Dairy allergy
* Presence of any serious medical conditions which might influence sleep i.e cardiovascular diseases, diabetes, cancer, respiratory disease, other than mild asthma)
* History of bariatric surgery
* Taking any kind of medication which might affect regular sleep
* Taking any type of medication which might affect appetite
* Participating in any kind of dietary and/or weight loss programs
* Taking antidepressants
* Substance or alcohol abuse
* Shift work
* Currently having to wake up at night to care for another person
* Suffering from and/or receiving treatment for mental health conditions or sleep apnoea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Sweet Taste Preference | 0-4 weeks
  Preference for sweetness will be assessed by providing participants with 5ml volumes of 5 sucrose solutions with concentrations 3%, 6%, 12%, 24% and 36% in random order. Preference for sweetness will be assessed by asking participants to rate the pleasantness of the solution on a VAS with anchors of 'not at all pleasant' and 'extremely pleasant'.
  To determine the preferred optimal sweetness, participants will be presented with pairs of 5 sucrose solutions and asked which solution they prefer. This will continue until the participants consistently choose a preference for a solution twice a row. A maximum of 10 trials will be conducted to assess preference. This assessment will be done fasted and fed state.
Sweet Taste Perception | 0-4 weeks
  Perception of sweetness will be assessed by providing participants with 5ml volumes of 5 sucrose solutions with concentrations 3%, 6%, 12%, 24% and 36% in random order. The perception of sweetness will be measured via visual analogue scale (VAS) to rate the sweetness of the solution with anchors of 'not at all sweet' and 'extremely sweet'.
Fat Taste Preference | 0-4 weeks
  Preference for fat taste will be assessed by providing participants with 5ml volumes 5 solutions with combinations with concentrations 3%, 6%, 12%, 24% and 36% fat (comprising skimmed milk and double cream mixes of different proportions) in random order. Preference for fat taste will be assessed by asking participants to rate pleasantness of the solution on a VAS with anchors of 'not at all' and 'extremely'.
  To determine the preferred optimal fat taste, participants will be presented with 5 pairs of milk and cream mix solutions and asked which solution they prefer. This will continue until the participants consistently choose a preference for one solution twice in a row. A maximum of 10 trials will be conducted to assess preference. This assessment will be done fasted and fed state.
Fat Taste Perception | 0-4 weeks
  Perception and preference for fat will be assessed by providing participants with 5ml volumes 5 solutions with combinations with concentrations 3%, 6%, 12%, 24% and 36% fat (comprising skimmed milk and double cream mixes of different proportions) in random order. The perception of fat will be measured via a visual analogue scale (VAS) to rate the creaminess of solution with anchors of 'not at all' and 'extremely'.

SECONDARY OUTCOMES:
Food preference - explicit liking | 0-4 weeks
  Changes in explicit liking measured by the Leeds Food Preference Questionnaire
  This assessment will be conducted in a fasted and post-prandial state.
  Scale range:
  Changes in explicit liking measured by the Leeds Food Preference Questionnaire.
  Scoring:
  The minimum score for VAS scale is 0 and maximum is 100. Scores are recorded and converted in to mean scores for high fat, low fat, sweet or savoury food types and different fat-taste combinations.
Food preference - explicit wanting | 0-4 weeks
  Changes in explicit wanting measured by the Leeds Food Preference Questionnaire
  This assessment will be conducted in a fasted and post-prandial state.
  Scale range:
  Changes in explicit wanting measured by the Leeds Food Preference Questionnaire.
  Scoring:
  The minimum score for VAS scale is 0 and maximum is 100. Scores are recorded and converted in to mean scores for high fat, low fat, sweet or savoury food types and different fat-taste combinations.
Food reward - implicit wanting | 0-4 weeks
  Changes in implicit wanting and food choice measured by the Leeds Food Preference Questionnaire
  This assessment will be conducted in a fasted and post-prandial state.
  Scale range:
  The computerized asessment where participants are presented with two images and they choose which they like.
  Scoring:
  Reaction time for each answer is recorded and converted in to mean scores for high fat, low fat, sweet or savoury food types and different fat-taste combinations.
Control of Eating Questionnaire - Craving control | 0-4 weeks
  Changes in craving control measured by the Control of Eating Questionnaire
  This assessment will be conducted in a fasted and post-prandial state.
  Scale range:
  The asessment includes a 20 items with a 10 point scale ranging from "not at all" to "extremely" and 1 item with free text answer.
  Scoring:
  The minimum score for VAS scale is 0 and maximum is 100. The sum of items were calculated and divided by number of items in the subscale.
Control of Eating Questionnaire - Craving for sweet | 0-4 weeks
  Changes in craving for sweet measured by the Control of Eating Questionnaire
  This assessment will be conducted in a fasted and post-prandial state.
  Scale range:
  The asessment includes a 20 items with a 10 point scale ranging from "not at all" to "extremely" and 1 item with free text answer.
  Scoring:
  The minimum score for VAS scale is 0 and maximum is 100. The sum of items were calculated and divided by number of items in the subscale.
Control of Eating Questionnaire - Craving for savoury | 0-4 weeks
  Changes in craving for savoury measured by the Control of Eating Questionnaire
  This assessment will be conducted in a fasted and post-prandial state.
  Scale range:
  The asessment includes a 20 items with a 10 point scale ranging from "not at all" to "extremely" and 1 item with free text answer.
  Scoring:
  The minimum score for VAS scale is 0 and maximum is 100. The sum of items were calculated and divided by number of items in the subscale.
Control of Eating Questionnaire - Positive mood | 0-4 weeks
  Changes in positive mood measured by the Control of Eating Questionnaire
  This assessment will be conducted in a fasted and post-prandial state.
  Scale range:
  The asessment includes a 20 items with a 10 point scale ranging from "not at all" to "extremely" and 1 item with free text answer.
  Scoring:
  The minimum score for VAS scale is 0 and maximum is 100. The sum of items were calculated and divided by number of items in the subscale. Higher the score indicates higher cravings.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gill, PhD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom